CLINICAL TRIAL: NCT00797069
Title: Comparison of Nutritional Products for People With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Bobbie Swearengin, Director Clinical Research, Abbott Nutrition
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BK20
Record Dates: First submitted 2008-11-23; First posted 2008-11-25 (Estimated); Last update posted 2010-07-30 (Estimated); Status verified 2010-03

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- standard nutritional product (Active Comparator): Standard nutritional product not specific for diabetes
  Interventions: Other: standard nutritional product (medical food)
- diabetes specific product (Active Comparator): Diabetes specific nutritional product
  Interventions: Other: nutritional product for diabetes (medical food)
- Experimental diabetes specific product (Experimental): Diabetes specific experimental nutritional product
  Interventions: Other: diabetes specific experimental nutritional product (medical food)

INTERVENTIONS:
Other: standard nutritional product (medical food) — once during crossover
  Arms: standard nutritional product
Other: nutritional product for diabetes (medical food) — once during crossover
  Arms: diabetes specific product
Other: diabetes specific experimental nutritional product (medical food) — once during crossover
  Arms: Experimental diabetes specific product

SUMMARY:
Compare the glycemic and insulinemic responses of a standard nutritional product with two diabetes-specific nutritional products in patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Subject states that he/she has type 2 diabetes (as evidenced by use of oral hypoglycemic medication for at least two months).
2. Subject is between 18 and 75 years of age, inclusive.
3. Subject is a male or a non-pregnant, non-lactating female, at least 6 weeks postpartum prior to screening visit.
4. If female is of childbearing potential, is practicing a method of birth control.
5. Subject's BMI is > 18.5 kg/m2 and < 35 kg/m2.
6. If on a chronic medication such as anti-hypertensive, lipid-lowering, thyroid medication or hormone therapy, subject has been on constant dosage for at least two months prior to screening visit.

Exclusion Criteria:

1. Subject uses exogenous insulin for glucose control.
2. Subject states that he/she has type 1 diabetes.
3. Subject states that he/she has a history of diabetic ketoacidosis.
4. Subject takes an alpha-glucosidase inhibitor.
5. Subject states that he/she has a current infection ; has had inpatient surgery, or corticosteroid treatment in the last 3 months or antibiotics in the last 3 weeks prior to screening visit.
6. Subject states that he/she has an active malignancy (excluding the following dermal malignancies: basal cell carcinoma, squamous cell carcinoma, carcinoma in-situ of the cervix).
7. Subject states that he/she has had a significant cardiovascular event ≤ six months prior to screening visit; or stated history of congestive heart failure.
8. Subject states that he/she has end stage organ failure or is status post organ transplant.
9. Subject states that he/she has a history of renal disease.
10. Subject states that he/she has current hepatic disease.
11. Subject states that he/she has a history of severe gastroparesis.
12. Subject states that he/she has a chronic, contagious, infectious disease, such as active tuberculosis, Hepatitis B or C, or HIV.
13. Subject has taken/is currently taking any herbals, dietary supplements, or medications, other than oral hypoglycemic medications, during the past four weeks prior to screening visit that could profoundly affect blood glucose.
14. Subject states that he/she has clotting or bleeding disorders.
15. Subject is known to be allergic or intolerant to any ingredient found in the study products.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2008-11; Primary Completion 2009-02 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
To compare the postprandial glycemic response of patients with type 2 diabetes consuming single servings of a standard liquid nutrition product and two diabetes-specific liquid nutrition products. | Three crossover periods

SECONDARY OUTCOMES:
To compare the postprandial insulinemic response of patients with type 2 diabetes consuming single servings of a standard liquid nutrition product and two diabetes-specific liquid nutrition products. | Three crossover periods

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Williams, MS, Study Chair — Abbott Nutrition
Locations (3):
- Spain (3):
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Miguel Servet, Zaragoza